CLINICAL TRIAL: NCT00560833
Title: A Multicenter, Randomized, Parallel-Group, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Four Different Doses of Org 50081 in the Treatment of Moderate to Severe Vasomotor Symptoms Associated With the Menopause
Brief Title: Dose-Finding Safety and Efficacy Trial of Org50081 (Esmirtazapine) in the Treatment of Vasomotor Symptoms (46101/P06459/MK-8265-012)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P06459; 46101 (Other: Organon Study Number); MK-8265-012 (Other: Merck Study Number); 2004-000469-36 (EudraCT Number)
Record Dates: First submitted 2007-11-16; First posted 2007-11-20 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Menopause; Vasomotor Symptoms
MeSH Terms: interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Participants receive placebo, encapsulated tablets, orally (PO), once daily (QD) for up to 12 weeks
  Interventions: Drug: Placebo
- Esmirtazapine 2.25 mg (Experimental): Participants receive esmirtazapine 2.25 mg, encapsulated tablets, PO, QD for up to 12 weeks
  Interventions: Drug: esmirtazapine
- Esmirtazapine 4.5 mg (Experimental): Participants receive esmirtazapine 4.5 mg, encapsulated tablets, PO, QD for up to 12 weeks
  Interventions: Drug: esmirtazapine
- Esmirtazapine 9 mg (Experimental): Participants receive esmirtazapine 9 mg, encapsulated tablets, PO, QD for up to 12 weeks
  Interventions: Drug: esmirtazapine
- Esmirtazapine 18 mg (Experimental): Participants receive esmirtazapine 18 mg, encapsulated tablets, PO, QD for up to 12 weeks
  Interventions: Drug: esmirtazapine

INTERVENTIONS:
Drug: esmirtazapine
  Other Names: Esmirtazapine maleate; SCH 900265; Org 50081
  Arms: Esmirtazapine 18 mg; Esmirtazapine 2.25 mg; Esmirtazapine 4.5 mg; Esmirtazapine 9 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The most direct treatment of vasomotor symptions (hot flushes) may be by means of 5-HT2A receptor antagonist. Mirtazapine is a potent blocker of 5-HT2A receptors and was found to be effective in reducing the number and intensity of hot flushes in preliminary trials. Also several Selective Serotonin Reuptake Inhibitors (SSRIs) and other similar compounds have been investigated to manage hot flushes, confirming the role of the serotonergic system. In the present trial, the efficacy and safety of four different doses of esmirtazapine compared to placebo was investigated in women with moderate to severe vasomotor symptoms associated with the menopause. The primary study hypothesis was that esmirtazapine would show superior efficacy to placebo.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women, defined as:
* 12 months of spontaneous amenorrhea;
* OR 6 months of spontaneous amenorrhea with serum Follicle Stimulating Hormone

(FSH) levels >40 mIU/mL;

* OR 6 weeks post surgical bilateral oophorectomy with or without hysterectomy.
* In case the menopausal status of a subject was unclear because of a hysterectomy, the serum FSH level had to be >40 mIU/mL. If the date of the last menstruation was not clear because of perimenopausal hormone use, then the subject had to have a serum FSH level >40 mIU/mL after completion of a washout period (see exclusion criteria below); be >= 40 and <= 65 years of age;
* have a body mass index (BMI) >= 18 and <= 32 kg/m^2;
* minimum of 7 moderate to severe hot flushes per day or 50 per week, as quantified from daily diary recordings during at least 7 days preceding randomization to trial medication;
* able to handle the electronic diary device after training and having at least 80% compliance on complete daily diary entries during the period prior to randomization;
* give voluntary written Informed Consent (IC) after the scope and nature of the investigation had been explained, before screening evaluations.

Exclusion Criteria:

* history or presence of any malignancy, except non-melanoma skin cancers
* any clinically unstable or uncontrolled renal, hepatic, endocrine,

respiratory, hematological, neurological, cardiovascular, or cerebrovascular disease that would put the subject at safety risk or mask measure of efficacy

* history of seizures or epilepsy; history or presence of clinically significant depression or other psychiatric disorder which, in the opinion of the investigator, might compromise or confound the participant's participation in the trial; abnormal clinically relevant vaginal bleeding
* any clinically relevant (opinion of investigator) abnormal finding during physical, gynecological and breast examination at screening; abnormal, clinically significant results of mammography. Mammography had to have been performed within the last 9 months prior to screening, otherwise it had to be done before inclusion into the trial. For non-US sites, if local laws or guidelines did not allow or advise such frequent mammograms, the documented local laws or guidelines were to be followed; abnormal cervical smear test results (corresponding to Pap III and higher, including Low-Grade Squamous Intraepithelial Lesion (LSIL), High-Grade Squamous Intraepithelial Lesion (HSIL), Cervical Intraepithelial Neoplasia (CIN) 1 and higher). A cervical smear had to have been performed within the last 9 months prior to screening, otherwise it had to be done before inclusion into the trial; hematological or biochemical values at screening outside the reference ranges considered clinically relevant in the opinion of the investigator
* high blood pressure (BP) (sitting systolic BP >170 mmHg and/or diastolic BP >100 mmHg)
* use of any drug product containing estrogens, progestins, androgens, or tibolone prior to screening (and up to and including randomization) within specified time frames

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 943 (Actual)
Dates: Start 2004-10-15 (Actual); Primary Completion 2006-01-15 (Actual); Study Completion 2006-01-15 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Birkhaeuser M, Bitzer J, Braat S, Ramos Y. Esmirtazapine treatment of postmenopausal vasomotor symptoms: two randomized controlled trials. Climacteric. 2019 Jun;22(3):312-322. doi: 10.1080/13697137.2018.1561664. Epub 2019 Feb 4. PMID 30712391
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P06459&kw=P06459&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 942 participants were randomly assigned to treatment in this study, however, one screened participant was given placebo treatment without a randomization assignment. This participant is included in the study placebo population.
Groups:
- Esmirtazapine 18mg: Participants receive esmirtazapine 18 mg, encapsulated tablets, PO, QD for up to 12 weeks
Period: Overall Study
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18mg
Started | 317 | 155 | 160 | 155 | 156
Treated | 317 (One participant was not randomized but was treated with placebo) | 154 (One participant was randomized but not treated) | 160 | 155 | 155 (One participant was randomized but not treated)
Completed | 273 | 129 | 121 | 124 | 114
Not Completed | 44 | 26 | 39 | 31 | 42
Not completed — Adverse Event | 16 | 10 | 25 | 23 | 35
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 22 | 9 | 6 | 4 | 4
Not completed — Participant uncooperative | 5 | 5 | 4 | 4 | 2
Not completed — Other | 1 | 1 | 3 | 0 | 0
Not completed — Never received drug | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received any study drug (placebo or esmertazapine), whether or not randomized.
Groups:
- Esmertazapine 18 mg: Participants receive esmertazapine 18 mg, encapsulated tablet, PO, QD for up to 12 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmertazapine 18 mg | Total
Number analyzed (Participants) | 317 | 154 | 160 | 155 | 155 | 941
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.0 (4.4) | 53.4 (4.4) | 54.1 (4.2) | 54.9 (4.8) | 54.1 (4.5) | 54.1 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 317 | 154 | 160 | 155 | 155 | 941
  Male | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Frequency of Vasomotor Symptoms (Frequency Score A) at Week 4
Description: Participants recorded the frequency of vasomotor symptoms (hot flushes) on an electronic diary card (LogPad®) on a daily basis during screening and treatment. Frequency score A was based on the number of moderate hot flushes + the number of severe hot flushes in one day. Baseline average was derived from, at most, 7 completely observed pre-treatment days. Weekly averages during treatment were calculated if at least 4 days with non-missing data were completely observed; if less than 4 days were completely observed, the averages of the previous week were carried forward (last observation carried forward, or LOCF). If the number of days observed in Week 1 were not sufficient, baseline values were carried forward.
Time Frame: Baseline and Week 4
Population: The intent-to-treat (ITT) population, defined as all randomized particpants having at least one recorded pre-baseline value of the number of moderate and severe hot flushes.
Measure: Mean (Standard Deviation); unit: Number of events
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18mg
Number analyzed (Participants) | 294 | 138 | 139 | 137 | 138
Number of events | -3.9 (4.2) | -5.6 (3.8) | -6.0 (3.6) | -6.0 (4.0) | -6.0 (4.4)
Statistical Analysis 1: Comparison: Placebo vs Esmirtazapine 2.25 mg; Test type: Superiority or Other; p < 0.01, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-2.3 to -0.4]
Statistical Analysis 2: Comparison: Placebo vs Esmirtazapine 4.5 mg; Test type: Superiority or Other; p < 0.01, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-3.1 to -1.2]
Statistical Analysis 3: Comparison: Placebo vs Esmirtazapine 9 mg; Test type: Superiority or Other; p < 0.01, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.9 to -1.0]
Statistical Analysis 4: Comparison: Placebo vs Esmirtazapine 18mg; Test type: Superiority or Other; p < 0.01, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.9 to -1.0]

2. Secondary Outcome: Change From Baseline in Vasomotor Symptoms Score Per Women's Health Questionnaire (WHQ) at Week 12
Description: The WHQ is a 36-item, user-friendly, and rapid way of assessing nine domains of physical and emotional health for mid-aged women. Participants self-administered the WHQ questionnaire; scoring is based on a 4-point scale as follows: 'Yes definitely=1', 'Yes sometimes=2', 'No not much=3' and 'No not at all=4'. Each score is transformed to a value '1' for scores '1' and '2' and to a value '0' for scores '3' and '4'. Vasomotor symptoms encompass Items 19 and 27 of the 36 total items. The transformed sums of items 19+27 are divided by 2 to get the score; therefore, the domain ranges from 0 to 1, where lower values are better.
Time Frame: Baseline and Week 12
Population: All participants receiving study drug with diary compliance adequate for this measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18mg
Number analyzed (Participants) | 282 | 136 | 135 | 133 | 136
Score on a scale
  Baseline | 0.984 (0.088) | 0.993 (0.060) | 0.985 (0.085) | 0.981 (0.114) | 0.985 (0.085)
  Change from baseline | -0.151 (0.329) | -0.235 (0.355) | -0.256 (0.355) | -0.256 (0.372) | -0.246 (0.385)

3. Primary Outcome: Change From Baseline in Average Daily Frequency of Vasomotor Symptoms (Frequency Score A) at Week 12
Description: Participants recorded the frequency of vasomotor symptoms (hot flushes) on a LogPad on a daily basis during screening and treatment. Frequency score A was based on the number of moderate hot flushes + the number of severe hot flushes in one day. Baseline average was derived from, at most, 7 completely observed pre-treatment days. Weekly averages during treatment were calculated if at least 4 days with non-missing data were completely observed; if less than 4 days were completely observed, the averages of the previous week were carried forward (last observation carried forward, or LOCF). If the number of days observed in Week 1 were not sufficient, baseline values were carried forward.
Time Frame: Baseline and Week 12
Population: The ITT population, defined as all randomized particpants having at least one recorded pre-baseline value of the number of moderate and severe hot flushes.
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18mg
Number analyzed (Participants) | 294 | 138 | 139 | 137 | 138
number of events | -4.9 (4.8) | -6.2 (5.1) | -6.7 (3.9) | -6.9 (4.4) | -6.5 (4.4)
Statistical Analysis 1: Comparison: Placebo vs Esmirtazapine 2.25 mg; Test type: Superiority or Other; p = 0.06, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-2.0 to 0.0]
Statistical Analysis 2: Comparison: Placebo vs Esmirtazapine 4.5 mg; Test type: Superiority or Other; p < 0.01, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-3.0 to -0.9]
Statistical Analysis 3: Comparison: Placebo vs Esmirtazapine 9 mg; Test type: Superiority or Other; p < 0.01, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.9 to -0.9]
Statistical Analysis 4: Comparison: Placebo vs Esmirtazapine 18mg; Test type: Superiority or Other; p < 0.01, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-2.6 to -0.5]

4. Primary Outcome: Change From Baseline in Average Daily Severity of Moderate/Severe Vasomotor Symptoms (Severity Score A) at Week 4
Description: Participants recorded the severity of hot flushes on a LogPad on a daily basis during screening and treatment. The severity of hot flushes was defined as: mild (sensation of heat without sweating); moderate (sensation of heat with sweating, able to continue activity); and severe (sensation of heat with sweating, causing cessation of activity). Severity score A was calculated as the number of moderate hot flushes x 2 + the number of severe hot flushes x 3, divided by the total number of moderate and severe hot flushes. If no hot flushes were experienced, this was to be recorded as 'no sensation of heat'. Baseline values were based on, at most, 7 completely observed pre-treatment days. If less than 4 days were completely observed during treatment, the averages of the previous week were carried forward (last observation carried forward, or LOCF). If the number of days observed in Week 1 were not sufficient, baseline values were carried forward.
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18mg
Number analyzed (Participants) | 294 | 138 | 139 | 137 | 138
score on a scale | -0.09 (0.23) | -0.11 (0.22) | -0.15 (0.25) | -0.16 (0.24) | -0.15 (0.24)
Statistical Analysis 1: Comparison: Placebo vs Esmirtazapine 2.25 mg; Test type: Superiority or Other; p = 0.62, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.09 to 0.03]
Statistical Analysis 2: Comparison: Placebo vs Esmirtazapine 4.5 mg; Test type: Superiority or Other; p = 0.02, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.12 to -0.01]
Statistical Analysis 3: Comparison: Placebo vs Esmirtazapine 9 mg; Test type: Superiority or Other; p = 0.01, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.13 to -0.01]
Statistical Analysis 4: Comparison: Placebo vs Esmirtazapine 18mg; Test type: Superiority or Other; p = 0.02, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.12 to -0.01]

5. Primary Outcome: Change From Baseline in Average Daily Severity of Moderate/Severe Vasomotor Symptoms (Severity Score A) at Week 12
Description: as for outcome 4
Time Frame: Baseline and Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18mg
Number analyzed (Participants) | 294 | 138 | 139 | 137 | 138
score on a scale | -0.12 (0.28) | -0.10 (0.27) | -0.15 (0.29) | -0.18 (0.26) | -0.17 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Esmirtazapine 2.25 mg; Test type: Superiority or Other; p = 1.0, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.06 to 0.07]
Statistical Analysis 2: Comparison: Placebo vs Esmirtazapine 4.5 mg; Test type: Superiority or Other; p = 0.72, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.09 to 0.04]
Statistical Analysis 3: Comparison: Placebo vs Esmirtazapine 9 mg; Test type: Superiority or Other; p = 0.13, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.12 to 0.01]
Statistical Analysis 4: Comparison: Placebo vs Esmirtazapine 18mg; Test type: Superiority or Other; p = 0.15, ANCOVA — Dunnet-adjusted from ANCOVA with factors for treatment and (pooled) center and a covariate for baseline value; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.12 to 0.01]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were collected up to 7 days after the last dose of study drug; serious adverse events were collected for up to 30 days after the last dose of study drug.
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18mg
Serious Adverse Events (participants affected / at risk) | 2/317 | 1/154 | 3/160 | 2/155 | 0/155
Other Adverse Events (participants affected / at risk) | 128/317 | 93/154 | 99/160 | 102/155 | 123/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=317) | Esmirtazapine 2.25 mg (N=154) | Esmirtazapine 4.5 mg (N=160) | Esmirtazapine 9 mg (N=155) | Esmirtazapine 18mg (N=155)
Appendicitis perforated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal lesion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=317) | Esmirtazapine 2.25 mg (N=154) | Esmirtazapine 4.5 mg (N=160) | Esmirtazapine 9 mg (N=155) | Esmirtazapine 18mg (N=155)
Abdominal distension (Gastrointestinal disorders) | 8 (8) | 5 (5) | 8 (12) | 3 (4) | 9 (10)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 9 (9) | 7 (7) | 18 (21) | 22 (23)
Nausea (Gastrointestinal disorders) | 17 (19) | 5 (5) | 5 (5) | 6 (7) | 5 (5)
Fatigue (General disorders) | 11 (12) | 19 (24) | 19 (20) | 19 (22) | 20 (23)
Oedema peripheral (General disorders) | 8 (10) | 9 (14) | 11 (11) | 7 (10) | 9 (9)
Nasopharyngitis (Infections and infestations) | 15 (16) | 10 (10) | 11 (11) | 11 (12) | 10 (11)
Weight increased (Investigations) | 18 (18) | 25 (25) | 24 (24) | 32 (33) | 45 (46)
Increased appetite (Metabolism and nutrition disorders) | 13 (14) | 12 (12) | 21 (21) | 14 (16) | 28 (29)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (17) | 5 (5) | 9 (10) | 14 (16) | 5 (5)
Dizziness (Nervous system disorders) | 12 (15) | 6 (10) | 12 (15) | 6 (7) | 14 (18)
Headache (Nervous system disorders) | 54 (74) | 11 (11) | 13 (18) | 14 (16) | 19 (26)
Lethargy (Nervous system disorders) | 1 (1) | 7 (7) | 14 (17) | 5 (6) | 4 (4)
Somnolence (Nervous system disorders) | 19 (20) | 33 (43) | 37 (49) | 44 (54) | 50 (63)
Insomnia (Psychiatric disorders) | 13 (18) | 6 (6) | 10 (10) | 6 (6) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less